CLINICAL TRIAL: NCT07220057
Title: Improving the Health of Americans Through Prevention and Management of Diabetes, Heart Disease and Stroke - Sustainable Culturally Adapted Nutrition (SCAN) Program
Brief Title: Sustainable Culturally Adapted Nutrition (SCAN) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Department of State Health Services (Other)
Responsible Party: Principal Investigator, William B Perkison, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-21-0180; HHS000353700001 (Other: Texas Department of State Health Services)
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sustainable Culturally Adapted Nutrition (SCAN) Program plus DPP plus Produce Delivery (Experimental): Participants will be a part of the Diabetes Prevention Program (DPP), and additionally, as a participant in the the SCAN program, will receive live online instructional video sessions and email links that provide additional training information. Participants will also receive produce delivery.
  Interventions: Behavioral: Live instructional video sessions; Behavioral: Links to educational videos; Behavioral: Diabetes Prevention Program (DPP); Behavioral: Produce Delivery
- Diabetes Prevention Program (DPP) plus Produce Delivery (Active Comparator): Participants will be a part of the Diabetes Prevention Program (DPP) and will also receive produce delivery.
  Interventions: Behavioral: Diabetes Prevention Program (DPP); Behavioral: Produce Delivery

INTERVENTIONS:
Behavioral: Live instructional video sessions — Three instructional live video sessions will be provided to participants via live videoconferencing. The session will describe fundamentals for preparing produce for cooking, healthy approaches to cooking foods, a review of serving sizes, reading labels, and different classes of health foods. The nutrition education is designed to promote healthy dietary patterns for all by empowering participants to navigate healthy eating through the lens of their own food and cultural experiences. By emphasizing culinary techniques over recipes, instructors can inspire adaptability of culturally familiar flavors and ingredients for a diverse range of ethnicities, abilities, and cooking equipment.
  Arms: Sustainable Culturally Adapted Nutrition (SCAN) Program plus DPP plus Produce Delivery
Behavioral: Links to educational videos — This online information will supplement and reinforce the information presented in the live instructional video sessions.
  Arms: Sustainable Culturally Adapted Nutrition (SCAN) Program plus DPP plus Produce Delivery
Behavioral: Diabetes Prevention Program (DPP) — The Diabetes Prevention Program (DPP) is a lifestyle change program intended to stop the onset of type 2 diabetes. The program involves Lifestyle Coaches, who help participants make and maintain the lifestyle changes that can help prevent type 2 diabetes. The Lifestyle Coaches share information about diabetes prevention, debunk fitness and health myths, and encourage fitness and healthy eating in regular group sessions. They also work with participants individually on personalized weight loss and exercise goals and action plans, using the group as a source of support and encouragement.
Behavioral: Produce Delivery — The investigators partnered with the Houston Food Bank (HFB) to offer up to 30 pounds of fresh produce twice per month to all DPP participants through a food prescription (Food Rx) program.

SUMMARY:
The purpose of the study is to determine the impact of an enhanced, food incentive program [called the sustainable culturally adapted nutrition (SCAN) program], which is integrated with the Diabetes Prevention Program (DPP) and a food prescription framework. The SCAN program aims is to improve participant adherence and the ability to make sustainable behavioral changes to reduce the chances of developing diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the DPP program conducted by First Mile
* Body Mass Index (BMI) ≥ 18
* fasting glucose of 100-126 milligrams per deciliter (mg/dL) and/or Hemoglobin A1C (HbA1C) 5.4%-6.5%

Exclusion Criteria:

* Withdrawal from the DPP program
* Participant opts to not specifically participate in the SCAN program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change in number of Diabetes Prevention Program (DPP) sessions attended | Baseline, at the end of the SCAN intervention (12 months after start of SCAN intervention)

SECONDARY OUTCOMES:
Change in Weight | Baseline, at the end of the SCAN intervention (12 months after start of SCAN intervention)
Change in calculated Body Mass Index (BMI) | Baseline, at the end of the SCAN intervention (12 months after start of SCAN intervention)
  BMI will be calculated as kg/m2.
Change in HbA1c level | Baseline, at the end of the SCAN intervention (12 months after start of SCAN intervention)
Low-Density Lipoprotein (LDL) level | Baseline, at the end of the SCAN intervention (12 months after start of SCAN intervention)
High-Density Lipoprotein (HDL) level | Baseline, at the end of the SCAN intervention (12 months after start of SCAN intervention)
Triglyceride level | Baseline, at the end of the SCAN intervention (12 months after start of SCAN intervention)

CONTACTS AND LOCATIONS:
Overall Officials: William Perkison, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No